CLINICAL TRIAL: NCT06725394
Title: Effect of Smartphone Addiction on Neck Disability During Pregnancy: the Mediating Role of Stress
Brief Title: Effect of Smartphone Addiction on Pregnancy
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Sena Dilek Aksoy, Principal Investigator, Kocaeli University
Other Study IDs: sdilek10
Record Dates: First submitted 2024-11-26; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2023-09

CONDITIONS: Smartphone Addiction; Neck Disability; Stress
Keywords: Mediation analysis; Pregnant women; Smartphone addiction; Neck disability; Stress
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group 1: Pregnant women
  Interventions: Other: Filling out the survey

INTERVENTIONS:
Other: Filling out the survey — Data were collected using an information form, the Smartphone Addiction Scale-Short Version (SAS-SV), the Perceived Stress Scale (PSS-10), and the Neck Disability Index (NDI).

SUMMARY:
This study will investigate the effect of smartphone addiction on neck disability during pregnancy and its mediating role on stress. The study will be conducted between September 2023 and April 2024. Data will be collected using the information form, Smartphone Addiction Scale-Short Version (SAS-SV), Perceived Stress Scale (PSS-10) and Neck Disability Index (NDI). Multiple regression and structural equation modeling will be used in the analysis of the data.

DETAILED DESCRIPTION:
Objective: After reviewing the relevant studies, we thought that smartphone addiction may negatively affect neck injury and perceived stress may play a mediating role in this relationship. In this context, our research questions are as follows:

* Do smartphone addiction and certain characteristics significantly predict stress in pregnant women?
* Do smartphone addiction and certain characteristics significantly predict neck injury in pregnant women?
* Does stress have a mediating effect on the relationship between smartphone addiction and neck injury in pregnant women? The research is a cross-sectional, analytical and screening study. The research will be conducted face-to-face with pregnant participants who apply to the pregnancy follow-up clinic of a public hospital and meet the research criteria and voluntarily participate in the research. Verbal and written consent will be obtained from all participants before data collection. The principles of the Declaration of Helsinki will be followed throughout the study. Data of the study will be collected using the Information Form, Smartphone Addiction Scale-Short Version (SAS-SV), Perceived Stress Scale-10 (PSS-10) and Neck Disability Index (NDI). Statistical analyses will be given as mean, standard deviation, median, minimum and maximum. T-tests will be used to compare categorical variables with scale scores, Pearson correlation to examine the relationship between scales and ANOVA to compare scale scores with three or more groups of categorical variables. Linear regression analysis will be used to examine the effects of SAS-SV scores and sociodemographic characteristics on PSS-10 and NDI. In addition, the mediating effect of PSS-10 on SAS-SV and NDI will be examined using a linear regression model. Analysis results will be considered significant at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18 and 49 years,
* With a gestational age of 20 weeks or more,
* No pregnancy complications,

Exclusion Criteria:

* Those with musculoskeletal system diseases (such as rheumatoid arthritis, ankylosing spondylitis, Scheuermann's disease, Ehlers-Danlos syndrome, spinal surgeries, nerve root compression, spondylolisthesis comorbidities)
* Those with diagnosed mental disorders

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women between the ages of 18-49
Sampling Method: Probability Sample
Enrollment: 428 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Filling out the survey | 30 minutes
  Filling out the tools used in the research

CONTACTS AND LOCATIONS:
Overall Officials: Sena Dilek Aksoy, Ph.D., Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No